CLINICAL TRIAL: NCT02933567
Title: CSC OnDemand: An Innovative Online Learning Platform for Implementing Coordinated Specialty Care
Acronym: CSCOnDemand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R44MH111283-01 (NIH)
Record Dates: First submitted 2016-09-24; First posted 2016-10-14 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CSC OnDemand Pilo (Experimental): Pilot Intervention
  Interventions: Other: CSC OnDemand

INTERVENTIONS:
Other: CSC OnDemand — CSC OnDemand is a multifaceted online learning product that includes four levels: 1) an online readiness tool and CSC Learning Hub; 2) dynamic multimedia core curriculum on first episode psychosis and CSC; 3) live faculty-led online courses; and 4) ongoing support, including an online community of practice to support peer-to-peer learning.

SUMMARY:
In response to the growing need for training on interventions to address first episode psychosis, the Center for Social Innovation (C4) has partnered with experts in Coordinated Specialty Care (CSC) to develop and test CSC OnDemand: An Innovative Online Learning Platform for Implementing Coordinated Specialty Care. The product builds on the findings of the Recovery After an Initial Schizophrenia Episode (RAISE) studies, funded by the National Institute of Mental Health (NIMH). RAISE examined team-based models of care for people early in the course of schizophrenia. Through a Fast Track Small Business Innovation Research (SBIR) grant, investigators will prototype, test, refine, and evaluate the impact of CSC OnDemand.

DETAILED DESCRIPTION:
Building on existing resources and the expertise of our faculty and advisors, we will develop CSC OnDemand, a multifaceted online learning product that includes four levels: 1) an online readiness tool and CSC Learning Hub; 2) dynamic multimedia core curriculum on first episode psychosis and CSC; 3) live faculty-led online courses; and 4) ongoing support, including an online community of practice to support peer-to-peer learning.

During Phases I and II of this Fast Track SBIR, we will prototype, pilot test, build out, and evaluate the product through a cluster randomized non-inferiority study comparing it with InPerson training.

Phase I will build a robust prototype of the online platform and test it with 15-20 providers from three sites. This Phase will explore feasibility, acceptability, and preliminary effectiveness of the product, and will examine which components of the online platform providers find most useful.

Based on our findings from Phase I, we will refine and fully build out the product to test in a larger randomized trial. Phase II will use a cluster randomized non-inferiority design to assess if OnDemand training (n = 20 sites) is comparable to InPerson training (n = 10 sites). Using a mixed-methods approach, we will examine provider (n = 150) outcomes (satisfaction; knowledge gains/retention; attitudes toward shared decision making) and client (n = 600) outcomes (work/school participation; engagement in CSC services; inpatient psychiatric hospitalizations).

The study is guided by the following specific aims:

Phase I AIM 1: To develop a prototype version of CSC OnDemand. AIM 2: To test the prototype online platform with a small sample of sites/providers to determine feasibility, acceptability, and preliminary effectiveness of the product.

Hypothesis: CSC OnDemand will show positive learning and satisfaction outcomes among providers, and findings will suggest the need for and feasibility of conducting a Phase II effectiveness trial.

Phase II AIM 1: To refine, expand, and finalize CSC OnDemand based on Phase I findings. AIM 2: To determine if the OnDemand training intervention is as successful as the InPerson intervention in increasing CSC providers knowledge and shared decision making (SDM). Hypothesis: Providers in the OnDemand condition will achieve increases in knowledge, SDM and satisfaction at post training and nine months that will be no more than .5 standard deviations less than the InPerson condition.

AIM 3: To determine if the OnDemand training intervention is as successful as the InPerson training in increasing participation in work or school, improving engagement in treatment, and decreasing relapse rates for participating clients.

Hypothesis: Clients being served by the providers in the OnDemand condition will have work/school participation rates, levels of engagement and rates of hospitalization nine months after admission that are no more than 10 percent higher (hospitalization) or lower (work/school, engagement) than clients served by providers in the InPerson condition.

ELIGIBILITY:
Inclusion Criteria: (providers in agencies)

* To be eligible, agencies will need to provide:

  1. direct care to individuals with early psychosis;
  2. administrative-level support for training and use of the CSC model;
  3. an entire treatment team that is willing to participate in this team-based intervention;
  4. contact information for direct service staff;
  5. support for the study, including a staff person to serve as a liaison to work with the research team;
  6. access to the Internet during the intervention period; and
  7. a willingness to provide data and participate in the evaluation.

Exclusion criteria:

1. Teams should not have previously received CSC training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Knowledge Test: Percentage of correct responses on a 50-item, complex multiple choice knowledge (effectiveness) test that is both discipline-specific and inclusive of all disciplines. | 2 weeks
  Participants will be tested on preliminary effectiveness of the CSC OnDemand tool.

SECONDARY OUTCOMES:
Satisfaction and Acceptability Survey: Level of satisfaction and acceptability with the CSC OnDemand tool as measured by quantitative and qualitative measures. | 2 weeks
  Participants will respond to satisfaction and acceptability questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olivet, MA, Principal Investigator — Center for Social Innovation
Locations (1):
- Center for Social Innovation, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes